CLINICAL TRIAL: NCT02186795
Title: Improvement in Total Hip Arthroplasty Patient Outcomes With Regional Anesthesia and Multimodal Analgesia: A Retrospective Analysis
Brief Title: Total Hip Arthroplasty Outcomes With Regional and Multimodal Analgesia
Acronym: THA
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Sylvia Wilson, Assistant Professor, Medical University of South Carolina
Other Study IDs: THA Retrospective Analysis
Record Dates: First submitted 2014-07-03; First posted 2014-07-10 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-06

CONDITIONS: Arthroplasty; Replacement, Hip; Arthritis
Keywords: Arthroplasty; Replacement, Hip
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lumbar plexus: Patients received a preoperative lumbar plexus nerve block (20 ml, ropivacaine 0.5%) for postoperative pain management with one to four multimodal oral pain medications (acetaminophen, celecoxib, oxycodone ER, gabapentin, pregabalin) administered preoperatively or in the first 48 hours postoperatively.
- Lumbar Epidural: Patients received a lumbar epidural preoperatively for postoperative pain management. Epidural infusions of ropivacaine 0.2% were initiated intraoperatively, administered until the morning of postoperative day 1, and titrated to patient comfort.

SUMMARY:
The goal of this retrospective chart review is to evaluate if the implementation of lumbar plexus block placement for postoperative pain and administration of multimodal oral analgesia have improved conditions in the postoperative period for patients undergoing total hip arthroplasty when compared to the placement of epidurals for postoperative pain management.

DETAILED DESCRIPTION:
Primary outcome: 48 hour opiate consumption in patients following THA. ' Secondary outcome: Time to first ambulation, assitstance needed with ambulation, opiate and regional related side effects, time to discharge orders.

ELIGIBILITY:
Inclusion Criteria:

1. Primary total hip arthroplasty, (identified by current procedural terminology (CPT) code 27130) and
2. Either a) Epidural or b) Lumbar plexus peripheral nerve block with the administration of multimodal medication after July 2012.

   -

   Exclusion Criteria:Exclusion criteria include THA Revision, ICU admission postoperatively, and dementia, not allowing pain score communication.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary total hip arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Wilson, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion criteria consisted of primary elective THA surgery with either (1) a lumbar epidural (n = 51) or (2) a lumbar plexus peripheral nerve block (n = 312) for postoperative analgaesia. Exclusion criteria were THA revision, traumatic fractures, nonelective surgery, general anaesthesia, and post-operative intensive care unit (ICU) admission.
Pre-assignment Details: Of the charts reviewed, 31 lumbar epidural and 153 lumbar plexus patients met inclusion criteria and were assigned a chronological number based on the date of their operation (Epidural 1-31; Lumbar plexus 1-153). These numbered lists were then randomised and data collected on the first 24 randomised patients for each block type.
Period: Overall Study
Arm/Group | Lumbar Plexus | Lumbar Epidural
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumbar Plexus | Lumbar Epidural | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (2.32) | 61.2 (2.55) | 61.65 (2.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 18 | 23 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Opiate Consumption
Description: Cumulative 48 Hours Opiate Consumption in Intravenous (IV) Morphine mg Equivalents (MME)
Time Frame: 48 hours postoperative
Measure: Mean (Standard Error); unit: IV MME
Arm/Group | Lumbar Plexus | Lumbar Epidural
Number analyzed (Participants) | 24 | 24
IV MME | 48.6 (5.21) | 53.9 (6.31)

ADVERSE EVENTS:
Time Frame: 48 hours after surgery or hospital discharge, whichever came first.
Arm/Group | Lumbar Plexus | Lumbar Epidural
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No